CLINICAL TRIAL: NCT02685501
Title: Menorrhagia, Dysmenorrhea and Iron Deficiency Among Young Women Soldiers
Brief Title: Menorrhagia, Dysmenorrhea and Iron Deficiency Among Young Women Soldiers and Effect on Activity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Shoshana Vilk, Prof. Shoshana Revel-Villk, Hadassah Medical Organization
Other Study IDs: Menorrhagia-HMO-CTIL
Record Dates: First submitted 2016-02-14; First posted 2016-02-18 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Menorrhagia; Dysmenorrhea; Iron Deficiency Anemia
MeSH Terms: conditions — Menorrhagia; Dysmenorrhea; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CBC, ferritin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Combat women soldiers: Women soldiers in combat units
  Interventions: Other: no intervention
- Non combat women soldiers: Women soldiers in non-combat units
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
As combat women soldiers are required to more intensive daily activity the investigators believe that the impact of menorrhagia, dysmenorrhea and its clinical consequence (as characterized by, anemia iron deficiency and reduced quality of life)) on personal performance will be more significant in combat women soldiers compared to non-combat women soldiers. Using cohorts from the same environment will enable the investigators to better study the effect of menorrhagia and dysmenorrhea eliminating other uncontrolled factors, such as nutrition. The study does not include any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women soldiers in the participating units

Exclusion Criteria:

* Lack of consent

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women soldiers
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Menorrhagia and dysmenorrhea | one year
  The prevalence of menorrhagia and dysmenorrhea and association with quality of life will be assessed

SECONDARY OUTCOMES:
Iron deficiency | one year
  The prevalence of iron deficiency and iron deficiency anemia will be assessed by laboratory tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided